CLINICAL TRIAL: NCT02131233
Title: A Phase III Multicenter, Double-Blind, Randomized, Active Comparator-Controlled Clinical Trial to Evaluate the Safety and Efficacy of Reformulated Raltegravir 1200 mg Once Daily Versus Raltegravir 400 mg Twice Daily, Each in Combination With TRUVADA™, in Treatment-Naïve HIV-1 Infected Subjects
Brief Title: Evaluation of the Safety and Efficacy of Reformulated Raltegravir (MK-0518) 1200 mg Once Daily in Combination With TRUVADA™ in Human Immunodeficiency Virus (HIV)-1 Infected, Treatment-Naive Participants (MK-0518-292)
Acronym: onceMRK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0518-292; 2013-001939-47 (EudraCT Number)
Record Dates: First submitted 2014-05-02; First posted 2014-05-06 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Reformulated Raltegravir (Experimental): Reformulated raltegravir 1200 mg (2x 600 mg tablets) orally once daily plus placebo to raltegravir 1 tablet orally twice daily plus TRUVADA™ orally once daily for 96 weeks
  Interventions: Drug: Reformulated Raltegravir; Drug: TRUVADA™; Drug: Placebo to Raltegravir
- Raltegravir (Active Comparator): Raltegravir 400 mg tablet orally twice daily plus placebo to reformulated raltegravir 2 tablets orally once daily plus TRUVADA™ orally once daily for 96 weeks
  Interventions: Drug: Raltegravir; Drug: TRUVADA™; Drug: Placebo to Reformulated Raltegravir

INTERVENTIONS:
Drug: Reformulated Raltegravir — Reformulated raltegravir 1200 mg (2x 600 mg tablets) orally once daily
  Arms: Reformulated Raltegravir
Drug: Raltegravir — Raltegravir 400 mg tablet orally twice daily
  Arms: Raltegravir
Drug: TRUVADA™ — Emtricitabine / tenofovir disoproxil fumarate 200 / 300 mg tablet administered once-daily with food (open-label)
Drug: Placebo to Reformulated Raltegravir — Placebo to reformulated raltegravir 2 tablets orally once daily
  Arms: Raltegravir
Drug: Placebo to Raltegravir — Placebo to raltegravir 1 tablet orally twice daily
  Arms: Reformulated Raltegravir

SUMMARY:
To evaluate the safety and efficacy of reformulated raltegravir (MK-0518) 1200 mg once daily in combination with TRUVADA™ versus raltegravir 400 mg twice daily in combination with TRUVADA™ in HIV-1 infected, treatment-naive participants. The primary hypothesis being tested is that reformulated raltegravir 1200 mg once-daily is non-inferior to raltegravir 400 mg twice-daily, each in combination therapy with TRUVADA™, as assessed by the proportion of participants achieving HIV-1 ribonucleic acid (RNA) <40 copies/mL at Week 48.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 positive
* Naïve to antiretroviral therapy including investigational antiretroviral agents
* Not of reproductive potential or, if of reproductive potential agrees to 1) true abstinence, or 2) use of an acceptable method of birth control during the study

Exclusion Criteria:

* Use of recreational or illicit drugs or has recent history of drug or alcohol abuse or dependence
* Has been treated for a viral infection other than HIV-1 (such as hepatitis B) with an agent that is active against HIV-1 including but not limited to adefovir, tenofovir, entecavir, emtricitabine, or lamivudine
* Has documented or known resistance to raltegravir, emtricitabine, and/or tenofovir before the first dose of study drug
* Has participated in a study with an investigational compound or device within 30 days or anticipates participating in such a study during this study
* Has used systemic immunosuppressive therapy or immune modulators within 30 days or is anticipated to need them during the study (short courses of corticosteroids are allowed)
* Requires or is anticipated to require any of the following prohibited medications while in the study: phenobarbital, phenytoin, rifampin, rifabutin, or calcium, magnesium and aluminum containing antacids, such as TUMS™, Maalox™ and Milk of Magnesia™
* Has significant hypersensitivity or other contraindication to any of the components of the study drugs
* Has current, active diagnosis of acute hepatitis due to any cause
* Is pregnant, breastfeeding, or expecting to conceive during the study
* Female participant expecting to donate eggs or male participant expecting to donate sperm during the study
* Is or has a family member (spouse or children) who is investigational staff or sponsor staff directly involved in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 802 (Actual)
Dates: Start 2014-05-23 (Actual); Primary Completion 2015-12-21 (Actual); Study Completion 2016-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Cahn P, Kaplan R, Sax PE, Squires K, Molina JM, Avihingsanon A, Ratanasuwan W, Rojas E, Rassool M, Bloch M, Vandekerckhove L, Ruane P, Yazdanpanah Y, Katlama C, Xu X, Rodgers A, East L, Wenning L, Rawlins S, Homony B, Sklar P, Nguyen BY, Leavitt R, Teppler H; ONCEMRK Study Group. Raltegravir 1200 mg once daily versus raltegravir 400 mg twice daily, with tenofovir disoproxil fumarate and emtricitabine, for previously untreated HIV-1 infection: a randomised, double-blind, parallel-group, phase 3, non-inferiority trial. Lancet HIV. 2017 Nov;4(11):e486-e494. doi: 10.1016/S2352-3018(17)30128-5. Epub 2017 Sep 11. PMID 28918877
- [Result] Cahn P, Sax PE, Squires K, Molina JM, Ratanasuwan W, Rassool M, Bloch M, Xu X, Zhou Y, Homony B, Hepler D, Teppler H, Hanna GJ, Nguyen BY, Greaves W; ONCEMRK Study Group. Raltegravir 1200 mg Once Daily vs 400 mg Twice Daily, With Emtricitabine and Tenofovir Disoproxil Fumarate, for Previously Untreated HIV-1 Infection: Week 96 Results From ONCEMRK, a Randomized, Double-Blind, Noninferiority Trial. J Acquir Immune Defic Syndr. 2018 Aug 15;78(5):589-598. doi: 10.1097/QAI.0000000000001723. PMID 29771789

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: These results stop at Week 96.
Period: Overall Study
Arm/Group | Reformulated Raltegravir | Raltegravir
Started | 533 (Enrolled participants) | 269 (Enrolled participants)
Treated | 531 | 266
Completed | 467 (Completed to Week 96) | 227 (Completed to Week 96)
Not Completed | 66 | 42
Not completed — Not Treated | 2 | 3
Not completed — Adverse Event | 7 | 6
Not completed — Death | 0 | 1
Not completed — Lack of Efficacy | 6 | 3
Not completed — Lost to Follow-up | 14 | 13
Not completed — Non-Compliance With Study Drug | 8 | 5
Not completed — Physician Decision | 7 | 0
Not completed — Pregnancy | 4 | 0
Not completed — Withdrawal by Subject | 18 | 11

BASELINE CHARACTERISTICS:
Population: All Treated Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Reformulated Raltegravir | Raltegravir | Total
Number analyzed (Participants) | 531 | 266 | 797
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.4 (10.3) | 36.9 (11.0) | 35.9 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 32 | 123
  Male | 440 | 234 | 674

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving <40 Copies/mL Human Immunodeficiency Virus-1 (HIV-1) Ribonucleic Acid (RNA) at Week 48
Description: From blood samples collected at week 48, HIV-1 RNA levels were determined by the Abbott RealTime HIV-1 Assay, which has a limit of reliable quantification (LoQ) of 40 copies/mL. The NC=F approach as defined by FDA "snapshot" approach was used as the primary approach to analysis where all missing data were treated as failures regardless of the reason.
Time Frame: Week 48
Population: All randomized participants who received at least one dose of study treatment
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Reformulated Raltegravir | Raltegravir
Number analyzed (Participants) | 531 | 266
Percentage of participants | 88.9 [85.9 to 91.4] | 88.3 [83.9 to 91.9]
Statistical Analysis 1: Comparison: Reformulated Raltegravir vs Raltegravir; The 95% Confidence Interval (CI) for the treatment differences in percent response were calculated using stratum-adjusted Mantel-Haenszel method with the difference weighted by the harmonic mean of sample size per arm for each stratum (screening HIV-1 RNA <=100,000 copies/mL or HIV-1 RNA >100,000 copies/mL); Test type: Non-Inferiority or Equivalence — Reformulated Raltegravir is concluded non-inferior to Raltegravir if the lower bound of the 95% CI for the difference in percent response is above -10 percentage points; Estimated Difference = 0.510, 95% CI 2-sided [-4.204 to 5.223] — Reformulated Raltegravir minus Raltegravir

2. Secondary Outcome: Percentage of Participants Achieving <40 Copies/mL Human Immunodeficiency Virus-1 (HIV-1) Ribonucleic Acid (RNA) at Week 96
Description: From blood samples collected at week 96, HIV-1 RNA levels were determined by the Abbott RealTime HIV-1 Assay, which has a limit of reliable quantification (LoQ) of 40 copies/mL. The NC=F approach as defined by FDA "snapshot" approach was used as the primary approach to analysis where all missing data were treated as failures regardless of the reason.
Time Frame: Week 96
Population: All randomized participants who received at least one dose of study treatment
Measure: Number; unit: Percentage of participants
Arm/Group | Reformulated Raltegravir | Raltegravir
Number analyzed (Participants) | 531 | 266
Percentage of participants | 81.5 [85.9 to 91.4] | 80.1 [83.9 to 91.9]
Statistical Analysis 1: Comparison: Reformulated Raltegravir vs Raltegravir; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Estimated Difference = 1.449, 95% CI 2-sided [-4.410 to 7.308] — Reformulated Raltegravir minus Raltegravir

3. Secondary Outcome: Change From Baseline in Cluster of Differentiation 4 (CD4) Cell Count at Week 48
Description: CD4 cells were counted from blood collected at baseline and week 48, and the change from baseline determined from week 48 minus baseline values.
Time Frame: Baseline and Week 48
Population: All randomized participants who received at least one dose of study treatment and have baseline data. The Observed Failure (OF) approach to handling missing values assumed baseline-carry-forward for all failures, and excluded other missing values.
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Reformulated Raltegravir | Raltegravir
Number analyzed (Participants) | 499 | 251
cells/mm^3 | 232.0 [214.6 to 249.4] | 234.1 [212.8 to 255.3]
Statistical Analysis 1: Comparison: Reformulated Raltegravir vs Raltegravir; The 95% CI for mean difference in CD4 change was based on t-distribution; Test type: Superiority or Other; Mean Difference (Final Values) = -2.1, 95% CI 2-sided [-30.9 to 26.7] — Reformulated Raltegravir minus Raltegravir

4. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 96
Description: CD4 cells were counted from blood collected at baseline and week 96, and the change from baseline determined from week 96 minus baseline values.
Time Frame: Baseline and Week 96
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Reformulated Raltegravir | Raltegravir
Number analyzed (Participants) | 482 | 235
cells/mm^3 | 261.6 [242.9 to 280.3] | 262.2 [236.4 to 288.0]
Statistical Analysis 1: Comparison: Reformulated Raltegravir vs Raltegravir; The 95% CI for mean difference in CD4 change was based on t-distribution; Test type: Superiority or Other; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-32.8 to 31.6] — Reformulated Raltegravir minus Raltegravir

5. Secondary Outcome: Percentage of Participants With an Adverse Event (AE) at Week 48
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE.
Time Frame: Up to Week 48
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Reformulated Raltegravir | Raltegravir
Number analyzed (Participants) | 531 | 266
Percentage of participants | 83.2 | 88.0

6. Secondary Outcome: Percentage of Participants With an AE After 96 Weeks of Treatment
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE.
Time Frame: Up to Week 98 (96 weeks of treatment + 2 weeks of follow up)
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Reformulated Raltegravir | Raltegravir
Number analyzed (Participants) | 531 | 266
Percentage of participants | 90.8 | 94.0

7. Secondary Outcome: Percentage of Participants With a Drug-Related AE at Week 48
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE. An investigator who is a qualified physician evaluated whether or not an AE was drug-related.
Time Frame: Up to Week 48
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Reformulated Raltegravir | Raltegravir
Number analyzed (Participants) | 531 | 266
Percentage of participants | 25.0 | 27.1

8. Secondary Outcome: Percentage of Participants With a Drug-Related AE After 96 Weeks of Treatment
Description: as for outcome 7
Time Frame: Up to Week 98 (96 weeks of treatment + 2 weeks of follow up)
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Reformulated Raltegravir | Raltegravir
Number analyzed (Participants) | 531 | 266
Percentage of participants | 26.4 | 28.6

9. Secondary Outcome: Percentage of Participants With a Serious Adverse Event (SAE) at Week 48
Description: A serious adverse event (SAE) is any AE occurring at any dose or during any use of Sponsor's product that does the following: results in death; is life threatening; results in persistent or significant disability/incapacity; results in or prolongs an existing inpatient hospitalization; is a congenital anomaly/birth defect; is a cancer; is associated with an overdose; is another important medical event.
Time Frame: Up to Week 48
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Reformulated Raltegravir | Raltegravir
Number analyzed (Participants) | 531 | 266
Percentage of participants | 6.2 | 9.4

10. Secondary Outcome: Percentage of Participants With a SAE After 96 Weeks of Treatment
Description: A SAE is any AE occurring at any dose or during any use of Sponsor's product that does the following: results in death; is life threatening; results in persistent or significant disability/incapacity; results in or prolongs an existing inpatient hospitalization; is a congenital anomaly/birth defect; is a cancer; is associated with an overdose; is another important medical event.
Time Frame: Up to Week 98 (96 weeks of treatment + 2 weeks of follow up)
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Reformulated Raltegravir | Raltegravir
Number analyzed (Participants) | 531 | 266
Percentage of participants | 9.6 | 15.8

11. Secondary Outcome: Percentage of Participants With a Serious and Drug-Related AE at Week 48
Description: A SAE is any AE occurring at any dose or during any use of Sponsor's product that does the following: results in death; is life threatening; results in persistent or significant disability/incapacity; results in or prolongs an existing inpatient hospitalization; is a congenital anomaly/birth defect; is a cancer; is associated with an overdose; is another important medical event. An investigator who is a qualified physician evaluated whether or not a SAE is drug-related.
Time Frame: Up to Week 48
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Reformulated Raltegravir | Raltegravir
Number analyzed (Participants) | 531 | 266
Percentage of participants | 0.2 | 0.8

12. Secondary Outcome: Percentage of Participants With a Serious and Drug-Related AE After 96 Weeks of Treatment
Description: as for outcome 11
Time Frame: Up to Week 98 (96 weeks of treatment + 2 weeks of follow up)
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Reformulated Raltegravir | Raltegravir
Number analyzed (Participants) | 531 | 266
Percentage of participants | 0.2 | 0.8

13. Secondary Outcome: Percentage of Participants Who Discontinued From Drug Therapy Due to an AE at Week 48
Description: as for outcome 6
Time Frame: Up to Week 48
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Reformulated Raltegravir | Raltegravir
Number analyzed (Participants) | 531 | 266
Percentage of participants | 1.1 | 2.3

14. Secondary Outcome: Percentage of Participants Who Discontinued From Drug Therapy Due to an AE up to Week 96
Description: as for outcome 6
Time Frame: Up to Week 96
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Reformulated Raltegravir | Raltegravir
Number analyzed (Participants) | 531 | 266
Percentage of participants | 1.3 | 2.3

ADVERSE EVENTS:
Time Frame: Up to Week 98 (96 weeks of treatment + 2 weeks of follow up)
Description: All randomized participants who received at least one dose of study treatment.
Groups:
- Raltegravir 1200 mg QD + Truvada: Reformulated raltegravir 1200 mg (2x 600 mg tablets) orally once daily plus placebo to raltegravir 1 tablet orally twice daily plus TRUVADA™ orally once daily for 96 weeks
- Raltegravir 400 mg BID + Truvada: Raltegravir 400 mg tablet orally twice daily plus placebo to reformulated raltegravir 2 tablets orally once daily plus TRUVADA™ orally once daily for 96 weeks
Arm/Group | Raltegravir 1200 mg QD + Truvada | Raltegravir 400 mg BID + Truvada
Serious Adverse Events (participants affected / at risk) | 51/531 | 42/266
Other Adverse Events (participants affected / at risk) | 375/531 | 184/266
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raltegravir 1200 mg QD + Truvada (N=531) | Raltegravir 400 mg BID + Truvada (N=266)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastrointestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Drug ineffective (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Acquired immunodeficiency syndrome (Infections and infestations) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 2 (2)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cerebral toxoplasmosis (Infections and infestations) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis C (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Lymphogranuloma venereum (Infections and infestations) | 0 (0) | 1 (2)
Meningitis tuberculous (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Perineal abscess (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Plasmodium vivax infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Proctitis chlamydial (Infections and infestations) | 1 (1) | 0 (0)
Proctitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Rectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 1 (1)
Syphilis (Infections and infestations) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma of salivary gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Immunoblastic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Facial paresis (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 4 (4) | 2 (2)
Emotional distress (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 2 (2) | 0 (0)
Schizophrenia (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Lymphocele (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raltegravir 1200 mg QD + Truvada (N=531) | Raltegravir 400 mg BID + Truvada (N=266)
Abdominal pain (Gastrointestinal disorders) | 46 (57) | 12 (15)
Diarrhoea (Gastrointestinal disorders) | 71 (82) | 34 (42)
Nausea (Gastrointestinal disorders) | 72 (88) | 34 (38)
Vomiting (Gastrointestinal disorders) | 42 (45) | 20 (24)
Fatigue (General disorders) | 40 (44) | 17 (19)
Influenza like illness (General disorders) | 14 (16) | 14 (19)
Pyrexia (General disorders) | 26 (30) | 15 (16)
Bronchitis (Infections and infestations) | 29 (32) | 14 (16)
Influenza (Infections and infestations) | 31 (41) | 18 (22)
Nasopharyngitis (Infections and infestations) | 65 (88) | 26 (35)
Syphilis (Infections and infestations) | 28 (30) | 19 (21)
Upper respiratory tract infection (Infections and infestations) | 67 (90) | 27 (37)
Accidental overdose (Injury, poisoning and procedural complications) | 29 (35) | 17 (25)
Blood creatine phosphokinase increased (Investigations) | 26 (31) | 18 (19)
Arthralgia (Musculoskeletal and connective tissue disorders) | 27 (32) | 7 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 39 (47) | 14 (15)
Dizziness (Nervous system disorders) | 39 (46) | 19 (20)
Headache (Nervous system disorders) | 84 (106) | 37 (45)
Depression (Psychiatric disorders) | 17 (19) | 15 (17)
Insomnia (Psychiatric disorders) | 31 (31) | 18 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 40 (48) | 17 (19)
Pruritus (Skin and subcutaneous tissue disorders) | 18 (21) | 17 (18)
Rash (Skin and subcutaneous tissue disorders) | 30 (35) | 13 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.